CLINICAL TRIAL: NCT02407054
Title: A Double-Blinded, Placebo-Controlled, Randomized Phase II Study of Enzalutamide With or Without the PI3 Kinase/mTOR Inhibitor LY3023414 in Men With Metastatic Castration Resistant Prostate Cancer
Brief Title: A Study of Enzalutamide and LY3023414 in Men With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Sarah Cannon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15798; I6A-MC-CBBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — LY3023414; enzalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD (Experimental): Participants received 200 milligrams (mg) LY3023414 orally twice daily (BID) during the initial week to assess pharmacokinetics (PK). Thereafter, participants received 200 mg of LY3023414 BID in combination with 160 mg of enzalutamide QD beginning Cycle 1 Day 1. A treatment cycle was defined as 28 days.
  Interventions: Drug: LY3023414; Drug: Enzalutamide
- Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD (Experimental): Participants received 200 mg LY3023414 orally BID in combination with 160 mg enzalutamide orally once daily (QD).
  Interventions: Drug: LY3023414; Drug: Enzalutamide
- Part B: Placebo + 160 mg Enzalutamide QD (Active Comparator): Participants received placebo in combination with 160 mg enzalutamide QD.
  Interventions: Drug: Enzalutamide; Drug: Placebo

INTERVENTIONS:
Drug: LY3023414 — Administered orally
  Arms: Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD; Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD
Drug: Enzalutamide — Administered orally
Drug: Placebo — Administered orally
  Arms: Part B: Placebo + 160 mg Enzalutamide QD

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of the study drug known as LY3023414 in combination with enzalutamide in men with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Metastatic disease documented by positive bone scan or metastatic lesions on computed tomography (CT) or magnetic resonance imaging (MRI) scan.
* Prostate cancer progression documented by PSA and/or radiographic progression according to prostate cancer working group 2 (PCWG2).
* Prior abiraterone treatment completed at least 4 weeks prior to cycle 1 day 1. Participants must have failed prior abiraterone treatment.
* Surgically or medically castrated, with testosterone levels of < 50 nanograms/deciliter.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
* Ability to swallow the study drugs whole.
* Adequate hematologic function.
* Adequate coagulation parameters, defined as international normalization ratio (INR) ≤ 2.
* Availability of tumor tissue from any time since diagnosis of prostate cancer disease. If no tumor samples are available the participant might still be eligible following discussion between the investigator and the medical monitor.

Exclusion Criteria:

* Prior cytotoxic chemotherapy, immunotherapy, a PI3K/AKT/mTOR agent (including TORC1 and TORC2 inhibitors), or RA 223 dichloride for the treatment of castration resistant prostate cancer (CRPC). Participants may have received docetaxel in the hormone-sensitive setting.
* Prior investigational new generation potent anti-androgen therapy (such as ARN 509).
* Prior treatment with enzalutamide.
* Pathological finding consistent with small cell carcinoma of the prostate.
* Prior systemic treatment with an azole drug (fluconazole, itraconazole) within 4 weeks of cycle 1 day 1.
* Known brain metastasis.
* History of (a) seizure or any condition that may predispose to seizure (prior cortical stroke or significant brain trauma); (b) loss of consciousness or transient ischemic attack within 12 months prior to day 1 of cycle 1.
* Uncontrolled hypertension (systolic blood pressure [BP] ≥ 160 millimeters of mercury [mmHg] or diastolic BP ≥ 95 mmHg).
* Have serious pre-existing medical conditions (at the discretion of the investigator).
* Have known acute or chronic leukemia or current hematologic malignancies that, in the judgment of the investigator and sponsor, may affect the interpretation of results.
* Have insulin-dependent diabetes mellitus. Participants with a type 2 diabetes mellitus are eligible if adequate control of blood glucose level is obtained by oral anti-diabetics as documented by hemoglobin A1c <7%.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g. ulcerative disease, uncontrolled nausea, vomiting, grade ≥2 diarrhea, and malabsorption syndrome).
* Have a history of New York Heart Association (NYHA) Class ≥3, QTc interval > 480 milliseconds (ms) on screening electrocardiogram (ECG) per Friderica's formula, unstable angina, or myocardial infarction (MI) in 6 months prior to study drug administration.
* Clinically significant electrolyte imbalance ≥ grade 2.
* Currently receiving treatment with therapeutic doses of warfarin sodium.
* Have initiated treatment with bisphosphonates or approved receptor activator of nuclear factor kappa-B ligand (RANK-L) targeted agents (e.g. denosumab) ≤28 days prior to day 1 of cycle 1.
* Concurrent serious infections requiring parenteral antibiotic therapy.
* Have a second primary malignancy that in the judgment of the investigator and medical monitor may affect the interpretation of results.
* Have an active, known fungal, bacterial, and/or known viral infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (36):
  - Urology Centers of Alabama, P.C., Homewood, Alabama
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Prostate Oncology Specialists, Marina del Rey, California
  - Sharp Memorial Hospital, San Diego, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Fort Wayne Oncology & Hematology, Fort Wayne, Indiana
  - Indiana Cancer Pavilion, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology/Hematology PA, Minneapolis, Minnesota
  - Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Garden State Urology, Morristown, New Jersey
  - Delaware Valley Urology, Voorhees Township, New Jersey
  - Associated Medical Professionals of NY, Syracuse, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Northwest Cancer Specialists PC, Tualatin, Oregon
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Univ of Pittsburgh Cancer Inst. (UPCI), Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Southwestern Medical Center - Dallas, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - US Oncology, The Woodlands, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Sweeney CJ, Percent IJ, Babu S, Cultrera JL, Mehlhaff BA, Goodman OB, Morris DS, Schnadig ID, Albany C, Shore ND, Sieber PR, Guba SC, Zhang W, Wacheck V, Donoho GP, Szpurka AM, Callies S, Lin BK, Bendell JC. Phase Ib/II Study of Enzalutamide with Samotolisib (LY3023414) or Placebo in Patients with Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2022 Jun 1;28(11):2237-2247. doi: 10.1158/1078-0432.CCR-21-2326. PMID 35363301
- See also: Click here for more information about this study: A Study of Enzalutamide and LY3023414 in Men With Prostate Cancer — http://www.lillytrialguide.com/EN-us/studies/cancer/cbbd

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who did not voluntarily withdraw, or who were not removed from the study due to adverse event (AE), non-compliance, or at their physician's decision were considered to be study completers.
Groups:
- Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD: Participants received 200 milligrams (mg) LY3023414 orally twice daily (BID) during initial week to assess pharmacokinetics (PK). Thereafter, participants received 200 mg of LY3023414 BID in combination with 160 mg of enzalutamide orally QD beginning Cycle 1 Day 1. A treatment cycle was defined as 28 days.
- Part B: Placebo + 160 mg Enzalutamide QD: Participants received placebo in combination with 160 mg enzalutamide orally QD.
Period: Overall Study
Arm/Group | Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD | Part B: Placebo + 160 mg Enzalutamide QD
Started | 13 | 65 | 64
Received at Least One Dose of Study Drug | 13 | 65 | 64
Completed | 6 | 47 | 57
Not Completed | 7 | 18 | 7
Not completed — Adverse Event | 1 | 4 | 1
Not completed — Non-compliance with Study | 0 | 2 | 1
Not completed — Physician Decision | 1 | 3 | 3
Not completed — Withdrawal by Subject | 5 | 9 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD: Participants received 200 mg LY3023414 orally every 12 hours (BID) during initial week to assess pharmacokinetics (PK). Thereafter, participants received 200 mg of LY3023414 BID in combination with 160 mg of enzalutamide orally QD beginning Cycle 1 Day 1. A treatment cycle was defined as 28 days.
- Total: Total of all reporting groups
Arm/Group | Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD | Part B: Placebo + 160 mg Enzalutamide QD | Total
Number analyzed (Participants) | 13 | 65 | 64 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (8.43) | 69.8 (8.30) | 70.9 (9.07) | 70.7 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 13 | 65 | 64 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 61 | 63 | 135
  Unknown or Not Reported | 2 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 6 | 4 | 12
  White | 11 | 53 | 55 | 119
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 65 | 64 | 142

OUTCOME MEASURES:

1. Primary Outcome: Part B: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization until the date of clinical (symptomatic or radiographic) and/or prostate specific antigen (PSA) disease progression per Prostate Cancer Clinical Trials Working Group (PCWG2) or death by any cause regardless of whether the participants withdraws from study drug or receives a subsequent anti-cancer therapy (as determined by the investigator). Participants who have not progressed or died at the time of assessment were censored at the time of the last date of assessment (tumor evaluation or PSA level).
Time Frame: Randomization to Measured Progressive Disease or Death from Any Cause (Up To 34 Months)
Population: All participants who received at least one dose of study drug in Part B. Per protocol, this analysis was planned for Part B only. Censored participants: Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD =19 and Part B: Placebo + 160 mg Enzalutamide QD =8.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD | Part B: Placebo + 160 mg Enzalutamide QD
Number analyzed (Participants) | 46 | 56
months | 3.78 [2.89 to 5.06] | 2.83 [2.27 to 3.22]
Statistical Analysis 1: Comparison: Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD vs Part B: Placebo + 160 mg Enzalutamide QD; Test type: Superiority; Hazard Ratio (HR) = 0.5871, 95% CI 2-sided [0.3967 to 0.8690]

2. Secondary Outcome: Part B: Time to Disease Progression (TTP)
Description: TTP was defined as time from randomization until the date of clinical (symptomatic or radiographic) and/or prostate specific antigen (PSA) disease progression per Prostate Cancer Clinical Trials Working Group (PCWG2).
Time Frame: Randomization to Objective Disease Progression (Up To 34 Months)
Population: All participants who received at least one dose of study drug in Part B. Per protocol, this analysis was planned for Part B only. Censored participants: Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD=32 and Part B: Placebo + 160 mg Enzalutamide QD=22.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD | Part B: Placebo + 160 mg Enzalutamide QD
Number analyzed (Participants) | 33 | 42
months | 5.06 [3.19 to 8.34] | 3.61 [2.86 to 4.70]
Statistical Analysis 1: Comparison: Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD vs Part B: Placebo + 160 mg Enzalutamide QD; Test type: Superiority; Hazard Ratio (HR) = 0.6515, 95% CI 2-sided [0.4123 to 1.0294]

3. Secondary Outcome: Part B: Percentage of Participants With Prostate Specific Antigen Response
Description: PSA response was defined as more than 50% and 90% reduction from baseline to lowest post baseline value. 95% Confidence Intervals are based on Fisher's Exact Method.
Time Frame: 12 Weeks
Population: All participants who received at least one dose of study drug in Part B. Per protocol, this analysis was planned for Part B only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD | Part B: Placebo + 160 mg Enzalutamide QD
Number analyzed (Participants) | 65 | 64
Percentage of participants
  50% PSA Response | 21.5 [12.3 to 33.5] | 25.0 [15.0 to 37.4]
  90% PSA Response | 7.6 [2.5 to 17.0] | 9.3 [3.5 to 19.3]

4. Secondary Outcome: Part A: Pharmacokinetic (PK): Area Under the Concentration-time Curve Over the Dosing Interval (AUCτ) of LY3023414
Description: PK: Area under the Concentration-time Curve Over the Dosing Interval (AUCτ) of LY3023414
  Time Frame:
  Part A LY3023414 200 mg: Day-1 pre-dose, 1.5, 3, and 6 hours post LY3023414 dose, Cycle 1 Day 1 pre-dose of LY3023414 and enzalutamide, and Part A Day 15 Pre-dose of LY3023414 and enzalutamide 1.5, 3, and 6 hours post LY3023414 dose;
Time Frame: Part A: 200 mg LY3023414 + 160 mg Enzalutamide: Cycle 1 Day 15 Pre-dose of LY3023414 and enzalutamide 1.5, 3, and 6 hours post LY3023414 dose
Population: All participants who received at least one dose of study drug and had evaluable PK data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Part A: 200 mg LY3023414: Participants received 200 mg LY3023414 orally every 12 hours (BID) during initial week to assess pharmacokinetics (PK).
- Part A: 200 mg LY3023414 BID + 160 mg Enzalutamide: Participants received 200 mg LY3023414 orally BID in combination with 160 mg enzalutamide orally once daily (QD) at the beginning Cycle 1 Day 1.
Arm/Group | Part A: 200 mg LY3023414 | Part A: 200 mg LY3023414 BID + 160 mg Enzalutamide
Number analyzed (Participants) | 11 | 8
nanogram*hour/milliliter (ng*h/mL) | 3230 (59) | 1820 (56)

5. Secondary Outcome: Part B: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 millimeter (mm), or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Second Measured Complete Response or Partial Response (Up To 34 Months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD | Part B: Placebo + 160 mg Enzalutamide QD
Number analyzed (Participants) | 65 | 64
percentage of participants | 4.6 [1.0 to 12.9] | 4.6 [1.0 to 13.1]

ADVERSE EVENTS:
Time Frame: Baseline Up To 5 Years
Description: All participants who received at least one dose of study drug.
Arm/Group | Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD | Part B: Placebo + 160 mg Enzalutamide QD
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/65 | 3/64
Serious Adverse Events (participants affected / at risk) | 5/13 | 13/65 | 12/64
Other Adverse Events (participants affected / at risk) | 13/13 | 64/65 | 63/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD (N=13) | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD (N=65) | Part B: Placebo + 160 mg Enzalutamide QD (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 200 mg LY3023414 BID + 160 mg of Enzalutamide QD (N=13) | Part B: 200 mg LY3023414 BID + 160 mg Enzalutamide QD (N=65) | Part B: Placebo + 160 mg Enzalutamide QD (N=64)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 11 (29) | 18 (34)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 1 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1) | 2 (3)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Ocular rosacea (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 1 (3) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 3 (5) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (5) | 6 (7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Anal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 11 (12) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 7 (17) | 40 (68) | 10 (12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 7 (7) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 4 (5) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 38 (58) | 25 (32)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 3 (3) | 3 (5) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 9 (10) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (12) | 18 (24) | 6 (12)
Asthenia (General disorders) | 3 (4) | 8 (9) | 4 (4)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (5) | 1 (1) | 2 (2)
Chills (General disorders) | 2 (2) | 5 (5) | 2 (2)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (11) | 41 (64) | 36 (45)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 3 (5) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 7 (7) | 5 (6)
Pain (General disorders) | 1 (1) | 0 (0) | 3 (5)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 3 (4)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (4) | 6 (10) | 6 (7)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 5 (8) | 5 (7)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (4) | 1 (2)
Blood creatinine increased (Investigations) | 1 (2) | 5 (8) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance (Investigations) | 1 (2) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 11 (17) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 20 (25) | 14 (14)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 8 (9) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 6 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (10) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 9 (12) | 18 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 14 (19) | 17 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 6 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (7) | 9 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 7 (7) | 8 (12)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 12 (13) | 6 (8)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 9 (9) | 5 (5)
Headache (Nervous system disorders) | 4 (6) | 3 (4) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 6 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 6 (7)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (3) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (3) | 5 (9) | 5 (5)
Proteinuria (Renal and urinary disorders) | 0 (0) | 6 (14) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (4)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 5 (5) | 4 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (9) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 1 (1)
Skin maceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 6 (6) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 6 (8) | 8 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-02-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02407054/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02407054/SAP_001.pdf